CLINICAL TRIAL: NCT07305610
Title: INFLUENCE OF SELECTED POSITIONS ON HIP ABDUCTORS STRENGTH AND ACTIVATION IN PATELLOFEMORAL PAIN SYNDROME IN MALES
Acronym: PFPS
Status: Not yet recruiting | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Gouda Mohamed, Dr, Ahram Canadian University
Other Study IDs: Cairo University
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Patellofemoral Pain (PFPS)
Keywords: Hip Abductors; Muscle Strength; Muscle Activity; Side-lying; Standing
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PFPS Group: Subjects with unilateral PFPS diagnosed by an orthopedist; age 18-35 years; normal BMI
- Control Group: Healthy individuals without knee pain; age 18-35 years; normal BMI

SUMMARY:
The study aims to explore the effect of body position (side-lying versus standing) on hip abductors muscle strength and activation in individuals with and without PFPS and then to compare these measures between the two groups in each position

DETAILED DESCRIPTION:
A cross-sectional comparative study involving 44 subjects (22 subjects with PFPS and 22 healthy controls), aged 18-35 years. The study will measure hip abductor muscle strength (Peak torque, Maximal total work) using the Biodex Isokinetic System 4 PRO and muscle activity (%MVC) of the gluteus medius, gluteus maximus, and tensor fascia lata using Surface EMG (Noraxon Ultium EMG). Measurements will be taken in both standing and side-lying positions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years; Normal BMI; Subjects in the PFPS group diagnosed with unilateral PFPS by an orthopedist; Healthy individuals without knee pain (for the control group)

Exclusion Criteria:

* History of lower limb surgery; Any neurological disorders; Musculoskeletal disorders affecting the lower limb; Additional sources of anterior knee pain (tendonitis, Osgood-Schlatter, bursitis, etc.); Any inflammatory diseases

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males
Study Population: 44 subjects, divided into 22 subjects with PFPS and 22 healthy controls, recruited from the outpatient clinics and staff/students of Ahram Canadian University
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Muscle activity (%MVC) of the gluteus medius, gluteus maximus, and tensor fascia lata | During the assessment procedure (single time point)
  using SEMG
Peak torque (Nm) of hip abductors muscles | During the assessment procedure (single time point)
  using isokinetic

SECONDARY OUTCOMES:
Maximal total work (J) during concentric and eccentric contractions | During the assessment procedure (single time point)
  Using Isokinetic
The Arabic Version of the Kujala Score (Anterior Knee Pain Scale) | Baseline/Pre-assessment
  A questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: mohamed gouda mohamed, bachelor of physical therapy, Study Chair — Teaching assistant, Department of Physiotherapy, Department of Physical Therapy for Musculoskeletal Disorders and its Surgery, Faculty of Physical Therapy, Ahram Canadian University, Giza, Egypt
Locations (1):
- Ahram Canadian University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
no specific reason

REFERENCES:
- [Background] de Castro MP, Sanchotene CG, Costa GV, Lopes CMS, Hubert M, de Brito Fontana H, Ruschel C. Comparison between side-lying and standing positions for hip abductor strength assessment. J Bodyw Mov Ther. 2022 Apr;30:181-186. doi: 10.1016/j.jbmt.2022.02.011. Epub 2022 Feb 12. PMID 35500969